CLINICAL TRIAL: NCT01756599
Title: Multi-centre Prospective Cohort of Childhood Leukaemia: Determinants of Health and Quality of Life of the Patients After Treatment for an Acute Leukaemia During Childhood or Adolescence - LEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-A00984-39; 2012-27 (Other: AP HM)
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Leukaemia During Childhood or Adolescence
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- leukaemia during childhood or adolescence (Experimental)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples

SUMMARY:
Regular advances in cancer treatment have dramatically improved the prognosis of children and adolescents with acute leukemia (AL), raising with a great acuity the problem of the late physical side effects, social integration, quality of life of the patients and their family as well as identification of the determinants of these outcomes. Large nationwide and international cohorts developed in general population (I4C, EPIC ELF…) are restricted to the study of childhood cancers occurrence. In addition, the national registries (French, European) of childhood cancers are designed to evaluate incidence and mortality, but not to produce individual detailed data on the follow-up and outcome of these children. Answering these questions supposes a comprehensive multidisciplinary approach resting on prospective cohorts of cancer survivors, specifically exploring the outcome of these children. These cohorts allow to identify prognostic factors of the health condition and social integration, and to propose adapted strategies of follow-up. The Childhood Cancer Survivor Study (CCSS), which remains the most important study, only concerns the North-American populations and rests on a self-reported follow-up assessment. In France, the LEA study, initiated in 2004 could answer some of these questions, but the representativeness and the size of the population (study initially limited to two areas PACA-Corsica and Lorraine) remain insufficient to study uncommon events. Similar approaches are conducted in Europe trough the broad collaborative Pancare network, to which the LEA program is associated.

ELIGIBILITY:
Inclusion Criteria:

* Respect for the criteria of inclusion in the troop;
* 24-month-old Survivor of recoil(drop) with regard to(compared with) the diagnosis for the Leukaemia Aiguës Myéloblastiques (LAM) and Leukaemia Aiguës Lymphoblastiques ( LAL) transplanted in 1st complete forgiveness; or in 48 months of recoil(drop) with regard to(compared with) the diagnosis for the LAL not transplanted in first complete forgiveness;
* Having given his(her,its) agreement to participate in the study;
* Authorized to participate in the study by the parents(relatives) or the legal representatives, for any minor subject; in the particular case of a minor(miner) become major during the follow-up, a grown-up consent will be collected(taken in).

Exclusion Criteria:

* Non compliance with the criteria of inclusion beforehand quoted,
* Initial Treatment(Processing) realized except 9 participating centers, even in case of moving in in the geographical zones covered by these centers during the phase of treatment(processing) or in the course of follow-up.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2900 (Estimated)
Dates: Start 2012-12; Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
the data (medical, socio-economic, behavioral, environmental…) of the medium and long-term outcome of a cohort of patients treated for childhood acute leukemia | 10 years

SECONDARY OUTCOMES:
The impact of the mortality / survival of this troop of patients, remote of the treatment of the leukaemia of the childhood. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille; pascal AUQUIER, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Oudin C, Berbis J, Bertrand Y, Vercasson C, Thomas F, Chastagner P, Ducassou S, Kanold J, Tabone MD, Paillard C, Poiree M, Plantaz D, Dalle JH, Gandemer V, Thouvenin S, Sirvent N, Saultier P, Beliard S, Leverger G, Baruchel A, Auquier P, Pannier B, Michel G. Prevalence and characteristics of metabolic syndrome in adults from the French childhood leukemia survivors' cohort: a comparison with controls from the French population. Haematologica. 2018 Apr;103(4):645-654. doi: 10.3324/haematol.2017.176123. Epub 2018 Jan 19. PMID 29351982
- [Derived] Saultier P, Auquier P, Bertrand Y, Vercasson C, Oudin C, Contet A, Plantaz D, Poiree M, Ducassou S, Kanold J, Tabone MD, Dalle JH, Lutz P, Gandemer V, Sirvent N, Thouvenin S, Berbis J, Chambost H, Baruchel A, Leverger G, Michel G. Metabolic syndrome in long-term survivors of childhood acute leukemia treated without hematopoietic stem cell transplantation: an L.E.A. study. Haematologica. 2016 Dec;101(12):1603-1610. doi: 10.3324/haematol.2016.148908. Epub 2016 Aug 11. PMID 27515247
- [Derived] Oudin C, Auquier P, Bertrand Y, Chastagner P, Kanold J, Poiree M, Thouvenin S, Ducassou S, Plantaz D, Tabone MD, Dalle JH, Gandemer V, Lutz P, Sirvent A, Villes V, Barlogis V, Baruchel A, Leverger G, Berbis J, Michel G. Late thyroid complications in survivors of childhood acute leukemia. An L.E.A. study. Haematologica. 2016 Jun;101(6):747-56. doi: 10.3324/haematol.2015.140053. Epub 2016 Mar 11. PMID 26969082